CLINICAL TRIAL: NCT05377385
Title: Evaluation of the Usability and Effect on the Metabolic Control of the Omnipod DASH Insulin Administration System in Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Evaluation of the Omnipod DASH in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/018
Record Dates: First submitted 2022-05-02; First posted 2022-05-17 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 1; Children; Metabolic Control; Patient Satisfaction
Keywords: Type 1 diabetes mellitus; child; insulin administration; Omnipod DASH; usability; metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Children and adolescents with type 1 diabetes mellitus who started in 2021 in the Jessa Hospital with the Omnipod DASH insulin administration device.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire about usability of the Omnipod DASH insulin administration system

SUMMARY:
In this study the usability of the Omnipod DASH insulin administration system is evaluated prospectively by two questionnaires. The effect on the metabolic control is evaluated retrospectively by analysis of data from the medical records of the patients.

DETAILED DESCRIPTION:
In the study the usability of the Omnipod DASH (= insulin patch pump) is evaluated prospectively by two questionnaires. The first questionnaire concerns practical items on the application of the pump (e.g. Is it easy to fill to pod?), the wearing of the pump (e.g. Is it comfortable to wear the pump?) and the comparison with insulin administration with insulin pens or other insulin pumps (e.g. is it less painful to administrate insulin by the Omnipod DASH pump). The second questionnaire asks for possible problems that the patients experienced during the wearing of the pump (e.g. did you experience an allergic skin reaction). The questions are formulated to be answered by a 5-point likert scale.

The metabolic control is studied retrospectively from data extracted from the medical records, i.e. the results of the determination of HbA1c and the results from continuous glucose monitoring (CGM) at the start, and after 2, 4 and 6 months of the wearing of the Omnipod DASH insulin pump.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with type 1 diabetes mellitus
* Patients who started in 2021 with the Omnipod DASH insulin administration system in the Jessa Hospital

Exclusion Criteria:

* Children and adolescents without type 1 diabetes mellitus
* Children and adolescents with type 1 diabetes treated with insulin pens or other insulin pumps

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with type 1 diabetes mellitus who started in 2021 in the Jessa Hospital with the Omnipod DASH insulin administration system
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Usability of and problems encountered with the Omnipod Dash insulin administration system | Through study completion, an average of 6 months
  Usability of and problems encountered with the Omnipod Dash insulin administration system is evaluated by 2 home made questionnaire evaluated by a 5 point Likert scale. The first questionnaire includes 3 questions about the application of the pod (e.g. it is easy to place the pod), 7 questions about the wearing of the pod (e.g. the pod doesn't hinder me during sleeping) and 11 questions comparing insulin administration with insulin pens (e.g. insulin administration with the pod is more discrete). The second questionnaire includes 9 questions about possible problems with the Omnipod DASH insulin administration system (e.g. I developped an allergic skin reaction).

SECONDARY OUTCOMES:
Metabolic control of type 1 diabetes mellitus | Before and during the first 6 months of wearing the Omnipod Dash insulin administration system
  Metabolic control of the type 1 diabetes mellitus measured by HbA1c levels and results from continuous glucose measurement data (e.g. time in range, time below range, time above range).

CONTACTS AND LOCATIONS:
Overall Officials: Guy Massa, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No